CLINICAL TRIAL: NCT05088382
Title: Period Tracker at Home Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1339
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Menstrual Cycles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LH Urine Test — Test for the qualitative measurement of LH in urine

SUMMARY:
This study will assess the usability of a Period Tracker product when used by lay users in their own homes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 45 years
* Menstrual cycles are 21-60 days long
* Seeking to predict when her next period will start
* Seeking to give informed consent and comply with the investigational procedures
* Has a compatible iPhone with internet access that they are willing to use for the study (iPhone 7+ and iOS 13 and above)

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Used Clearblue® me (Period Tracker app), Persona Contraception Monitor or Clearblue Advanced Fertility Monitor within the last six months
* Currently or previously employed by SPD, Abbott, Alere, Unipath, P&G or affiliates
* Has an immediate* relative currently or previously (within past 5 years) employed by SPD, Abbott, Alere, Unipath or P&G, or affiliates
* Is a qualified or trainee healthcare professional (HCP)
* Has professional experience of using dipstick type tests or lateral flow devices
* Using any treatment which may affect the menstrual cycle (e.g. contraceptive pill)
* Using hormone replacement medications containing LH or hCG (e.g. Pregnyl®)
* Is currently seeking to conceive
* Has been diagnosed with polycystic ovarian syndrome (PCOS)
* Has PCOS symptoms e.g. very irregular cycles, hirsutism *Immediate relatives are defined as parents, children, siblings or partner/spouse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females are the intended user of this product
Study Population: Women between the ages of 18 to 45 represent the intended user of the product
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Usability of the Period Tracker device when used at home | 28 days (approximately 1 menstrual cycle)
  Number of users scoring 3 or less on a 7 point Likert scale for various questions related to usability of the Period Tracker device after use at home

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Boxer, Principal Investigator — SPD Development Company; Raniero Zazzeroni, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom